CLINICAL TRIAL: NCT02604641
Title: Assessment of the Impact of a Coenzyme Q10 Supplementation on the Skin: Randomised, Double-blind, Placebo-controlled Pilot Study
Brief Title: Assessment of the Impact of a Coenzyme Q10 Supplementation on the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Collaborators: Valens Int. d.o.o., Slovenija (Industry); Institute of Nutrition, Slovenia (Nutris) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Q10 01-2014
Record Dates: First submitted 2015-11-04; First posted 2015-11-13 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Wrinkles; Ageing; Photoprotection
Keywords: skin rejuvenation; anti-ageing effects; minimal erythema dose; dermis structure; physiological skin condition; wrinkling; dry skin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): 0 mg CoQ10 daily
  Interventions: Dietary Supplement: Placebo group
- Quvital LD group (Active Comparator): 50 mg CoQ10 daily
  Interventions: Dietary Supplement: Quvital LD group
- Quvital HD group (Active Comparator): 150 mg CoQ10 daily
  Interventions: Dietary Supplement: Quvital HD group

INTERVENTIONS:
Dietary Supplement: Placebo group — Subjects will take 5 mL of placebo syrup (0 mg CoQ10/day) once per day for 12 weeks.
  Arms: Placebo group
Dietary Supplement: Quvital LD group — Subjects will take 5 mL of LD syrup (50 mg CoQ10/day) once per day for 12 weeks.
  Arms: Quvital LD group
Dietary Supplement: Quvital HD group — Subjects will take 5 mL of LD syrup (150 mg CoQ10/day) once per day for 12 weeks.
  Arms: Quvital HD group

SUMMARY:
Objective of the study is to determine the influence of dietary supplementation with coenzyme Q10 (CoQ10) on skin conditions. 33 healthy female subjects will be randomly assigned to a placebo group, a low-dose (LD) group receiving 50 mg CoQ10/day and a high-dose group (HD) receiving 150 mg CoQ10/day (11 subjects per group). A water-soluble form of CoQ10 with improved bioavailability (Quvital syrup with Q10vital®, Valens Int. d.o.o., Slovenia) will be used. Various skin parameters will be evaluated before the supplementation (the baseline), after 6 and after 12 weeks of supplementation. To evaluate the photoprotective potential of CoQ10 the minimal erythema dose (MED) will be determined before (the baseline) and after 12 weeks of the supplementation.

DETAILED DESCRIPTION:
Objective of the study is to determine the influence of dietary supplementation of CoQ10 in form of water-soluble Q10vital® on skin conditions. 33 healthy female subjects will be randomly assigned to a placebo group, a low-dose (LD) group receiving 50 mg CoQ10/day and a high-dose group (HD) receiving 150 mg CoQ10/day (11 subjects per group). A water-soluble form of CoQ10 with improved bioavailability (Quvital syrup with Q10vital®, Valens Int. d.o.o., Slovenia) will be used. The placebo or CoQ10 will be administered in the form of a syrup; all subjects will consume 5 mL of syrup daily for 12 weeks. The photoprotective potential of CoQ10 will be evaluated with a determination of the minimal erythema dose (MED) before (the baseline) and after 12 weeks of the supplementation. Other skin parameters will be evaluated before supplementation (the baseline), after 6 and after 12 weeks of supplementation. Comparison will be done as the mean of the individual ratios. The differences between the before-after condition will be analyzed with the statistical test of analysis of variance. In case of failure to find homogeneity in the variances the nonparametric ANOVA, the Willcoxon test, will be used. The results will be expressed as mean ± standard error for each group with a significance level of 0.05 for all the statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Signs of skin aging (mimic wrinkles/ poor skin tone/ visual dryness),
* Photoaged skin on the face,
* Expression of mimic wrinkles,
* Phototype II and III.

Exclusion Criteria:

* Allergy to ingredients of tested products
* High blood cholesterol and use of cholesterol-lowering medicines,
* Diagnosed diabetes
* Thyroid disease
* Inflammatory skin diseases,
* Regular use of dietary supplements 6 months or less before start of the study,
* Invasive rejuvenation treatments (botox injections, hyaluronic acid fillers, needle rollers, needle mesotherapy, etc.) 6 months or less prior to start of the study,
* Non-invasive rejuvenation treatments (radiofrequency, electrotherapy, ultrasound therapy, no-needle mesotherapy, etc.) 6 months or less prior to start of the study,
* The use of cosmetic products containing coenzyme Q10 6 months or less prior to start of the study,
* Gluteal hyperpigmentation,
* Expected sunbathing (also in solariums) within the study period.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Improvement of photoprotective function of the skin | after 12 weeks of the supplementation
  Minimal erythema dose (MED) of the skin will be determined. Skin on gluteal part of the body will be exposed to 10 different doses of UVB light and 24 hours after exposure MED will be determined.Higher MED indicates better photoprotective function of the skin.

SECONDARY OUTCOMES:
Reduction of the area of the periorbital facial wrinkles | after 6 and after 12 weeks of the supplementation
  Area of selected periorbital wrinkles will be quantitatively assessed using CSI programme.
Reduction of the volume of the periorbital facial wrinkles | after 6 and after 12 weeks of the supplementation
  Volume of selected periorbital wrinkles will be quantitatively assessed using CSI programme.
Reduction of wrinkles at different face areas | after 6 and after 12 weeks of the supplementation
  Expert assessment of wrinkles at different face areas (periorbital, frontal, glabelar, nasolabial areas etc.) will be done according to Lemperle Wrinkle assessment scale.
Improvement of the dermis structure | after 6 and after 12 weeks of the supplementation
  Ultrasound (US) images of the dermis will be taken and intensity of the dermis determined. Higher intensity of the dermis US images indicates improvement of the collagen and elastin network.
An increase of the dermis thickness | after 6 and 12 weeks of the supplementation
  Dermis thickness will be measured with ultrasound imaging of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Janko Zmitek, PhD, Study Chair — VIST - Faculty of Applied Sciences; Katja Zmitek, PhD, Study Director — VIST - Faculty of Applied Sciences; Liljana Mervic, PhD, Study Chair — UL MF; Tina Tina Pogačnik, BSc, Principal Investigator — VIST - Faculty of Applied Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Scientific paper with results of the study (Zmitek et al. 2016. The effect of dietary intake of coenzyme Q10 on skin parameters and condition: Results of a randomised, placebo-controlled, double-blind study; Biofactors. 43(1):132-140) — http://onlinelibrary.wiley.com/doi/10.1002/biof.1316/abstract